CLINICAL TRIAL: NCT00886912
Title: Prevention of Acute Mountain Sickness (AMS) by Intermittent Hypoxic Training
Brief Title: Training in Hypoxia to Prevent Acute Mountain Sickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Medical Clinic, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S-160/2008
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2009-04

CONDITIONS: Acute Mountain Sickness; Healthy
Keywords: mountain sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxia (Active Comparator): training in simulated altitude
  Interventions: Other: hypoxia
- Normoxia (Placebo Comparator): training under normoxic conditions
  Interventions: Other: normoxia

INTERVENTIONS:
Other: hypoxia — training in simulated altitude in a hypoxic chamber (normobaric hypoxia)
  Arms: Hypoxia
Other: normoxia — training under normoxic conditions
  Arms: Normoxia

SUMMARY:
Some studies suggest that high-altitude related illnesses - like acute mountain sickness - could be prevented by acclimatisation, reached at low altitude using training in simulated altitude. The purpose of this study is to determine whether training in hypoxia is suitable to prevent acute mountain sickness.

DETAILED DESCRIPTION:
In a three week-period, healthy probands undergo 3 times a week a bicycle ergometer training in simulated altitude followed by 1 week passive exposure at simulated low altitude. 5 days after last exposure, a field study starts performing a rapid ascent to the Capanna Regina Margherita (4559m). Acute mountain sickness is assessed by established scoring systems.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoker
* endurance training min. 2x/week

Exclusion Criteria:

* any diseases
* previous exposure to altitudes higher than 2000m (last 6 weeks)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute mountain sickness | after 20 hours at 4559m

SECONDARY OUTCOMES:
Severity of acute mountain sickness | after 20 hours at 4559m

CONTACTS AND LOCATIONS:
Overall Officials: Kai Schommer, MD, Principal Investigator — Departement of Sports Medicine, University of Heidelberg
Locations (1):
- Departement of Sports Medicine, University of Heidelberg, Heidelberg, Germany